CLINICAL TRIAL: NCT06304896
Title: Colchicine Versus Beta-blockers, Angiotensin-converting Enzyme Inhibitors, and Statins for Prevention of Chemotherapy-Induced Cardiomyopathy
Acronym: BASiC-CIC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arab Contractors Medical Centre (Other)
Responsible Party: Principal Investigator, Eslam Abbas, MBChB, MSc, Dr., Arab Contractors Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: #18240343
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chemotherapy Induced Systolic Dysfunction
MeSH Terms: interventions — Carvedilol; Ramipril; Rosuvastatin Calcium; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Cardioprotective Group (CPG) (Active Comparator): 50 patients will receive a low-dose Beta-blockers in the form of Carvedilol 6.25 mg PO twice daily, a low-dose ACE inhibitors in the form of Ramipril 2.5 mg PO once daily, and a statin in the form of rosuvastatin 20 mg oral tablets.
  Interventions: Drug: Carvedilol; Drug: Ramipril; Drug: Rosuvastatin
- The Immunomodulatory Group (IMG) (Active Comparator): 50 patients will receive Colchicine 0.6 PO once daily.
  Interventions: Drug: Colchicine
- The Placebo Control Group (PCG) (Placebo Comparator): 50 patients will receive a placebo as a control group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — Carvedilol 6.25 mg oral tablets. Prescribed: Twice daily PO with 200 mL of water.
  Other Names: Carvid; Coreg
  Arms: The Cardioprotective Group (CPG)
Drug: Ramipril — Ramipril 2.5 mg oral capsules. Prescribed: Once daily PO with 200 mL of water.
  Other Names: Tritace; Altace
  Arms: The Cardioprotective Group (CPG)
Drug: Rosuvastatin — Rosuvastatin 20 mg oral tablets. Prescribed: Once daily PO with 200 mL of water.
  Other Names: Crestor
  Arms: The Cardioprotective Group (CPG)
Drug: Colchicine — Colchicine 0.6 mg oral tablets/capsules. Prescribed: Once daily PO with 200 mL of water.
  Other Names: Colcrys; Mitigare
  Arms: The Immunomodulatory Group (IMG)
Drug: Placebo — Placebo oral capsules. Prescribed: Once daily PO with 200 mL of water.
  Arms: The Placebo Control Group (PCG)

SUMMARY:
BASiC-CIC Trial is a multicenter, double-blinded, randomized, placebo-controlled clinical trial to investigate whether repurposing colchicine or a combination of beta-blockers, angiotensin-converting enzyme (ACE) inhibitors, and statins will be effective as a prophylactic treatment for the prevention of chemotherapy-induced cardiomyopathy, reduction of major adverse cardiovascular events, and all-cause mortality.

DETAILED DESCRIPTION:
The 2021 European Society of Cardiology (ESC) guidelines recommend that the treatment with angiotensin-converting enzyme inhibitors (ACEi) and a beta-blocker (preferably carvedilol) should be considered in cancer patients developing left ventricle systolic dysfunction, defined as a 10% or more decrease in left ventricular ejection fraction (LVEF) from baseline value or a value lower than 50%, during anthracycline chemotherapy. This statement has a class of recommendation of II with a level of evidence B, which means that the weight of evidence/opinion is in favor of the usefulness of these treatments. The statement recommends starting the dual treatment after echocardiographic evidence of cardiac affection. Therefore, whether pre-treatment with these dual cardio-protective agents will protect the patient's heart from the toxic effects of the chemotherapeutic intervention is unclear.

Additionally, The 2022 ACC/AHA/HFSA American guidelines recommend that in asymptomatic patients with cancer therapy-related cardiomyopathy (ejection fraction<50%), angiotensin-receptor blocker (ARBs)and beta-blockers are reasonable to prevent progression to heart failure and improve cardiac function. The statement also recommends starting the dual treatment after echocardiographic evidence of cardiac affection. However, these guidelines state that in patients at risk of cancer therapy-related cardiomyopathy, initiation of beta blockers and ACEi/ARB for the primary prevention of drug-induced cardiomyopathy is of uncertain benefit and further clinical research is an unmet need. Accordingly, the effectiveness of preemptive use of ACEi-ARB and/or selected beta-blockers (such as carvedilol and nebivolol) in reducing the risk of cancer therapy-related cardiomyopathy has been investigated in a number of small clinical trials, with conflicting findings. Additionally, statins have pleiotropic therapeutic effects that range from endothelial stabilization to suppression of inflammation. However, its role in decreasing disease morbidity (repeated hospitalization) in established chronic heart failure is also uncertain.

On the other hand, colchicine is an immunomodulator that accumulates in the white blood cells and affects them in a variety of ways including decreasing motility, mobilization, and adhesion. Generally, colchicine appears to inhibit multiple proinflammatory mechanisms, while enabling increased levels of anti-inflammatory mediators. In a randomized trial involving patients with chronic coronary disease, the risk of cardiovascular events was significantly lower among those who received 0.5 mg of colchicine once daily than among those who received a placebo. Accordingly, colchicine can reduce the risk of cardiovascular events in patients with chronic coronary artery disease, but its efficacy in improving the functional status in patients with established chronic heart failure is also uncertain. While the use of this immunomodulatory agent in established heart failure is uncertain, its effectiveness in the prophylactic reduction of chemotherapy-induced cardiomyopathy in patients with normal pre-treatment ejection fraction has not been investigated.

Accordingly, 150 enrolled cancer patients who are candidates for guideline-directed anthracycline-based chemotherapy with or without the anti-HER2 trastuzumab at the time of presentation, will undergo the following:

* General and Local cardiac examination.
* CBC.
* Chemistry Panel including KFTs, LFTs.
* Serum electrolytes levels.
* Baseline resting surface 12 leads ECG followed by serial recording (monthly for a total of 6 months).
* Baseline Echocardiography followed by serial imaging every 2 months for a total of 6 months.
* Baseline serum BNP test/NT-proBNP followed by serial testing every 2 months for a total of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to performing study procedures.
* A cancer patient who is a candidate for a guideline-directed, anthracycline-based chemotherapy with or without the anti-HER2 trastuzumab.
* Baseline LVEF ≥ 50% without evident structural heart disease by pre-treatment echocardiographic examination.

Exclusion Criteria:

* Critically ill Cancer patients who are admitted to ICU.
* Ischemic cardiomyopathy with LVEF ≤ 50%.
* Dilated cardiomyopathy with LVEF ≤ 50%.
* Advanced valvular heart disease (severe valvular affection in the form of stenosis or regurgitation).
* Systolic BP < 90 mmHg or diastolic BP < 60 mmHg.
* Liver cell failure.
* End-stage chronic kidney disease on regular dialysis.
* Pregnancy.
* Lactation.
* Chronic muscle diseases such as dermatomyositis, polymyositis, or muscular dystrophy.
* Acute trauma or burns within 2 weeks.
* History of allergy to the implemented drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-induced cardiomyopathy | 6 months
  An identification of a drop in the LVEF using echocardiography more than or equal to 10% from the baseline at the time of presentation and/or a decline of the LVEF less than 50%.
Chemotherapy-induced cardiomyopathy | 6 months
  An identification of at least one value of serum NT-proBNP over 125 pg/mL in patients less than 75 years of age, or 450pg/mL in patients more than 75 years of age.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events | 6 months
  The non-fatal major cardiovascular adverse events include:
  * Non-fatal myocardial infarction.
  * Non-fatal stroke.
  * Hospitalization due to unstable angina.
  * Hospitalization due to serious arrhythmias.
  * Hospitalization due to heart failure.
All-Cause Mortality | 6 months
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Eslam Abbas, MBChB, MSc, Principal Investigator — Arab Contractors Medical Centre
Locations (1):
- Arab Contractors Medical Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun X, Duan J, Gong C, Feng Y, Hu J, Gu R, Xu B. Colchicine Ameliorates Dilated Cardiomyopathy Via SIRT2-Mediated Suppression of NLRP3 Inflammasome Activation. J Am Heart Assoc. 2022 Jul 5;11(13):e025266. doi: 10.1161/JAHA.122.025266. Epub 2022 Jun 29. PMID 35766262
- [Background] Zhang FS, He QZ, Qin CH, Little PJ, Weng JP, Xu SW. Therapeutic potential of colchicine in cardiovascular medicine: a pharmacological review. Acta Pharmacol Sin. 2022 Sep;43(9):2173-2190. doi: 10.1038/s41401-021-00835-w. Epub 2022 Jan 19. PMID 35046517
- [Background] Kuo MC, Chang SJ, Hsieh MC. Colchicine Significantly Reduces Incident Cancer in Gout Male Patients: A 12-Year Cohort Study. Medicine (Baltimore). 2015 Dec;94(50):e1570. doi: 10.1097/MD.0000000000001570. PMID 26683907
- [Background] Zhang T, Chen W, Jiang X, Liu L, Wei K, Du H, Wang H, Li J. Anticancer effects and underlying mechanism of Colchicine on human gastric cancer cell lines in vitro and in vivo. Biosci Rep. 2019 Jan 15;39(1):BSR20181802. doi: 10.1042/BSR20181802. Print 2019 Jan 31. PMID 30429232
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Bosch X, Rovira M, Sitges M, Domenech A, Ortiz-Perez JT, de Caralt TM, Morales-Ruiz M, Perea RJ, Monzo M, Esteve J. Enalapril and carvedilol for preventing chemotherapy-induced left ventricular systolic dysfunction in patients with malignant hemopathies: the OVERCOME trial (preventiOn of left Ventricular dysfunction with Enalapril and caRvedilol in patients submitted to intensive ChemOtherapy for the treatment of Malignant hEmopathies). J Am Coll Cardiol. 2013 Jun 11;61(23):2355-62. doi: 10.1016/j.jacc.2013.02.072. Epub 2013 Apr 10. PMID 23583763
- [Background] Golwala H. Enalapril/carvedilol for prevention of chemotherapy-induced heart failure: an end to the problem. J Am Coll Cardiol. 2013 Dec 24;62(25):2450-2451. doi: 10.1016/j.jacc.2013.06.059. Epub 2013 Sep 4. No abstract available. PMID 24013049
- [Background] Spallarossa P, Guerrini M, Arboscello E, Sicbaldi V. Enalapril and carvedilol for preventing chemotherapy-induced left ventricular systolic dysfunction. J Am Coll Cardiol. 2013 Dec 24;62(25):2451-2452. doi: 10.1016/j.jacc.2013.07.077. Epub 2013 Sep 4. No abstract available. PMID 24013048
- [Background] Smiseth OA, Edvardsen T, Skulstad H. Cardioprotection during chemotherapy: need for faster transfer of knowledge from cardiology to oncology and role for a cardio-oncologist. J Am Coll Cardiol. 2013 Jun 11;61(23):2363-4. doi: 10.1016/j.jacc.2013.02.073. Epub 2013 Apr 10. No abstract available. PMID 23583243
- [Background] Guglin M, Krischer J, Tamura R, Fink A, Bello-Matricaria L, McCaskill-Stevens W, Munster PN. Randomized Trial of Lisinopril Versus Carvedilol to Prevent Trastuzumab Cardiotoxicity in Patients With Breast Cancer. J Am Coll Cardiol. 2019 Jun 11;73(22):2859-2868. doi: 10.1016/j.jacc.2019.03.495. PMID 31171092
- [Background] Gulati G, Heck SL, Ree AH, Hoffmann P, Schulz-Menger J, Fagerland MW, Gravdehaug B, von Knobelsdorff-Brenkenhoff F, Bratland A, Storas TH, Hagve TA, Rosjo H, Steine K, Geisler J, Omland T. Prevention of cardiac dysfunction during adjuvant breast cancer therapy (PRADA): a 2 x 2 factorial, randomized, placebo-controlled, double-blind clinical trial of candesartan and metoprolol. Eur Heart J. 2016 Jun 1;37(21):1671-80. doi: 10.1093/eurheartj/ehw022. Epub 2016 Feb 21. PMID 26903532
- [Background] Kalay N, Basar E, Ozdogru I, Er O, Cetinkaya Y, Dogan A, Inanc T, Oguzhan A, Eryol NK, Topsakal R, Ergin A. Protective effects of carvedilol against anthracycline-induced cardiomyopathy. J Am Coll Cardiol. 2006 Dec 5;48(11):2258-62. doi: 10.1016/j.jacc.2006.07.052. Epub 2006 Nov 9. PMID 17161256
- [Background] Shah P, Garris R, Abboud R, Vasudev R, Patel H, Doshi R, Shamoon F, Bikkina M. Meta-Analysis Comparing Usefulness of Beta Blockers to Preserve Left Ventricular Function During Anthracycline Therapy. Am J Cardiol. 2019 Sep 1;124(5):789-794. doi: 10.1016/j.amjcard.2019.05.046. Epub 2019 Jun 6. PMID 31307662
- [Background] Wittayanukorn S, Qian J, Westrick SC, Billor N, Johnson B, Hansen RA. Prevention of Trastuzumab and Anthracycline-induced Cardiotoxicity Using Angiotensin-converting Enzyme Inhibitors or beta-blockers in Older Adults With Breast Cancer. Am J Clin Oncol. 2018 Sep;41(9):909-918. doi: 10.1097/COC.0000000000000389. PMID 28537988
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Deftereos S, Giannopoulos G, Panagopoulou V, Bouras G, Raisakis K, Kossyvakis C, Karageorgiou S, Papadimitriou C, Vastaki M, Kaoukis A, Angelidis C, Pagoni S, Pyrgakis V, Alexopoulos D, Manolis AS, Stefanadis C, Cleman MW. Anti-inflammatory treatment with colchicine in stable chronic heart failure: a prospective, randomized study. JACC Heart Fail. 2014 Apr;2(2):131-7. doi: 10.1016/j.jchf.2013.11.006. PMID 24720919
- [Background] Rogers JK, Jhund PS, Perez AC, Bohm M, Cleland JG, Gullestad L, Kjekshus J, van Veldhuisen DJ, Wikstrand J, Wedel H, McMurray JJ, Pocock SJ. Effect of rosuvastatin on repeat heart failure hospitalizations: the CORONA Trial (Controlled Rosuvastatin Multinational Trial in Heart Failure). JACC Heart Fail. 2014 Jun;2(3):289-97. doi: 10.1016/j.jchf.2013.12.007. Epub 2014 Apr 30. PMID 24952697
- [Background] Tavazzi L, Maggioni AP, Marchioli R, Barlera S, Franzosi MG, Latini R, Lucci D, Nicolosi GL, Porcu M, Tognoni G; Gissi-HF Investigators. Effect of rosuvastatin in patients with chronic heart failure (the GISSI-HF trial): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Oct 4;372(9645):1231-9. doi: 10.1016/S0140-6736(08)61240-4. Epub 2008 Aug 29. PMID 18757089
- [Background] van der Harst P, de Boer RA. Statins in the treatment of heart failure. Circ Heart Fail. 2010 May;3(3):462-4. doi: 10.1161/CIRCHEARTFAILURE.110.956342. No abstract available. PMID 20484198